CLINICAL TRIAL: NCT03810651
Title: Pilot Study of Pencil Beam Scanning Proton Beam Radiation Therapy in Patients With Renal Tumors
Brief Title: Pencil Beam Scanning in Patients With Renal Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-014386
Record Dates: First submitted 2019-01-15; First posted 2019-01-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Renal Tumor; Wilms Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell; Wilms Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal tumors (Other): Any patient with Wilms tumor or clear cell sarcoma of the kidney who would require radiation therapy as standard of care. Patients may receive an investigation drug for Wilms or CCSK given concurrently or within the first four weeks of the first fraction of proton therapy administration.
  Interventions: Other: Proton beam radiation using pencil beam scanning

INTERVENTIONS:
Other: Proton beam radiation using pencil beam scanning — Proton beam radiation using pencil beam scanning, characterized by Bragg peak dose deposition and high conformality of dose to target regions

SUMMARY:
This is a pilot study to assess acute toxicity in patients receiving flank irradiation using proton therapy for renal tumors.

DETAILED DESCRIPTION:
Patients with renal tumors including Wilms and clear cell sarcoma of the kidney (CCSK) are treated with multimodality therapy which may include surgery, chemotherapy, and radiation. While long-term disease control is excellent, these patients remain at risk for early and late toxicities partially from radiation. There have been no significant changes to traditional photon radiation fields, which encompass the post-operative bed, anterior abdomen, and vertebral body. Proton beam radiation using pencil beam scanning, which is characterized by Bragg peak dose deposition and high conformality of dose to target regions, is ideally suited to treat the retroperitoneum. This pilot study evaluates pencil beam scanning proton therapy (PBS-PT) to:

* result in low acute gastrointestinal toxicity in patients receiving radiation therapy for renal tumors as measured by laboratory evaluations, clinician-assessed, and patient reported health related quality of life outcomes
* decrease the duration of radiation therapy
* compare doses to organs at risk (OARs) using PBS-PT as compared to traditional photon fields

ELIGIBILITY:
Inclusion Criteria:

* Less than 30 years of age
* Diagnosis

  a. Any patient with Wilms tumor or clear cell sarcoma of the kidney who would require radiation therapy as standard of care including
  1. Any patient with favorable histology (FH), stage III disease
  2. Any patient with focal or diffuse anaplasia
  3. Any patient with CCSK
* The patient is a candidate for external beam radiotherapy based on standard of care for treatment of Wilms tumor or CCSK

Exclusion Criteria:

* Prior radiotherapy to the region of the study cancer
* Chemotherapy administered for diagnosis of Wilms tumor or CCSK
* Pregnant or breastfeeding

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-12-26 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any non-hematologic toxicity that occurs within 90 days following the start of proton therapy assessed with with NCI Common toxicity criteria (CTC Version 4.0) grades]. | 90 days
  Acute toxicity in patients receiving flank irradiation using proton therapy for renal tumors. Acute toxicity is defined as any non-hematologic toxicity that occurs within 90 days following the start of proton therapy. NCI Common toxicity criteria (CTC Version 4.0) grades will be employed. Individual category content listings are available to investigators at http://ctep.cancer.gov, with attention to the following System Organ Classes and CTCAE Adverse Events: General Disorders and Administration Site Conditions, Hepatobiliary Disorders, Blood and Lymphatic System Disorders, Gastrointestinal Disorders, Renal and Urinary Disorders, Injury, poisoning, or procedural complications, Metabolism and nutrition disorders, and Benign, Malignant, and Unspecified Neoplasms.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hill-Kayser, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No